CLINICAL TRIAL: NCT02910817
Title: Impact of Metformin on In Vitro Fertilization Outcomes in Overweight and Obese Polycystic Ovary Syndrome Women; A Quasi Experimental Study
Brief Title: Impact of Metformin on In Vitro Fertilization Outcomes in Overweight and Obese PCOS Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Lecturer of OBGYN in women health hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: obgy-115-2014
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin-treated group (Experimental): 51 overweight and obese women (BMI>24) with PCOS underwent their first fresh autologous IVF-embryo transfer cycle
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): A cohort of fifty-one cross matched PCOS women
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — The metformin-treated group received metformin (1000 mg per day) with the start of controlled ovarian stimulation (COH) until the day of the pregnancy check.
  Arms: Metformin-treated group
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
RCT to investigate whether metformin co-treatment would improve IVF outcomes in overweight and obese women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria restricted the patients to 39 years old with basal FSH < 10 IU/ml and normal TSH and prolacin.

Exclusion Criteria:

* Exclusion criteria were diabetes mellitus (excluded by GTT), renal or liver disease, associated male factor, documented tubal factor or pelvic adhesions, elevated 17 alfa hydroxyprogesterone level and FSH ≥10 IU/ml. We also excluded the women who started program or medications to reduce their weight and those who their partner has abnormal semen parameters according to the world health organization parameters (WHO, 2010)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total number of retrieved oocytes | Two weeks Metformin treatment

SECONDARY OUTCOMES:
Live birth rate | End of the pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Osama Abdalmageed, Principal Investigator — Women health center
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdalmageed OS, Farghaly TA, Abdelaleem AA, Abdelmagied AE, Ali MK, Abbas AM. Impact of Metformin on IVF Outcomes in Overweight and Obese Women With Polycystic Ovary Syndrome: A Randomized Double-Blind Controlled Trial. Reprod Sci. 2019 Oct;26(10):1336-1342. doi: 10.1177/1933719118765985. Epub 2018 Mar 25. PMID 29576001